CLINICAL TRIAL: NCT02358590
Title: The Effect of Health Action Process Approach Menu-Based Intervention on Vitamin D Adherence in Older Adult With Osteoporosis-Pilot Study
Brief Title: The Effect of Theory Menu-Based Intervention on Vitamin D Adherence in People With Osteoporosis-Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-026
Record Dates: First submitted 2015-01-28; First posted 2015-02-09 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAPA menu-based mini-video (Experimental): This group will watch mini-videos, which are multi-target menu-based interventions designed to deliver information about vitamin D adherence and its effect on osteoporosis
  Interventions: Behavioral: HAPA menu-based mini-video
- Standard care (Active Comparator): This group will be advised by the treating physician to take vitamin D
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: HAPA menu-based mini-video — The intervention will be a multi-target menu-based mini-videos designed to deliver information about vitamin D adherence and its effect on osteoporosis
  Arms: HAPA menu-based mini-video
Behavioral: Standard care — The treating physician will advice participants to take vitamin D
  Arms: Standard care

SUMMARY:
This pilot study evaluates the effect of theory menu-based mini-videos on vitamin D adherence in older adult with osteoporosis. Half of participants will watch the videos while the other half will receive usual care (treating physician advice).

DETAILED DESCRIPTION:
Osteoporosis is a common disease around the world. The morbidity and mortality attributed to osteoporosis is due to fracture. The evidence shows that vitamin D is effective in preventing osteoporotic fracture, however, adherence to vitamin D is low among people with osteoporosis (20%-60%). The Health Action Process Approach (HAPA) has been found useful to describe, explain, and predict changes in health behaviours in a variety of setting. Based on HAPA, mini-videos will be developed aiming to increase vitamin D adherence in people with osteoporosis. Mini-videos will address self-efficacy, outcome expectancy, risk perception and action and coping plan. This pilot study aims to evaluate the recruitment and participants' feedback about the mini-videos.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 50 years
* Have been diagnosed with primary osteoporosis
* Have low vitamin D level (less than 75nmol/L) recently (within the previous month)
* Fluent in English

Exclusion Criteria:

* Cognitive diseases
* Mal-absorption syndromes that may interfere with vitamin D absorption.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  The ability to recruit 20 participants
Feedback of participants about the mini-videos | 5 minutes
  A feedback form will be applied to participants within 5 minutes of watching the videos (the intervention)

SECONDARY OUTCOMES:
Serum level of vitamin D | after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Norma J. MacIntyre, PT, PhD, Study Chair — McMaster University
Locations (1):
- Osteoporosis Clininc affiliated to St. Joseph's Hospital, Hamilton, Ontario, Canada